CLINICAL TRIAL: NCT02101749
Title: Comparative Immune Response of Intradermal and Intramuscular Preparations of
Brief Title: Immune Response of Intradermal and Intramuscular Preparations of Inactive Seasonal Influenza Vaccine in Older Age Group.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Elderly Flu vaccine
Record Dates: First submitted 2013-12-28; First posted 2014-04-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Influenza, Human
Keywords: trivalent inactivated influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trivalent inactivated influenza (INTANZA) (Active Comparator): Intradermal injection
  Interventions: Biological: trivalent inactivated influenza
- trivalent inactivated influenza (VAXIGRIP) (Active Comparator): Intramuscle injection
  Interventions: Biological: trivalent inactivated influenza

INTERVENTIONS:
Biological: trivalent inactivated influenza — intradermal or intramuscular injection in the deltoid area.

SUMMARY:
This is a prospective, Open label randomized study. A total of 220 adults aged ≥ 60 years will be enrolled and randomized to one of 2 study arms:

1. Seasonal inactivated intradermal influenza vaccine (15 μg HA (hemagglutinin) per strain/ 0.1 ml dose) (group A - 110 participants)
2. Seasonal inactivated intramuscular influenza vaccine (15 μg HA per strain/ 0.5 ml dose) (group B - 110 participants) Groups A and B will receive the vaccine at day 1. Total follow up period is 60 days.

DETAILED DESCRIPTION:
The consent form will be reviewed and signed by the participant prior to any study-related procedures.

Potential study participants will be assessed based on inclusion and exclusion criteria. Screening procedures, which include taking medical history, vital signs, random blood for dextrostix and vaccination will be performed on day 1.

A total of 220 participants will be randomized into 2 study arms, of which each group of 110 vaccinees will receive either seasonal intradermal influenza vaccine [group A] or seasonal intramuscular influenza vaccine [group B]. The randomization route of vaccination will be kept in concealed envelope at the study site. It will be open after subject signed informed consent form and all inclusion exclusion criteria met for enrollment. Groups A and B will receive the vaccine at day 1. Clinical activities for groups A and B during each visit (total of 5 visits). Blood will be drawn and assayed (for baseline assessment) using HAI (hemagglutination inhibition assay) to the three influenza strains.

ELIGIBILITY:
Inclusion criteria:

* Male or female aged ≥ 60 years
* Healthy and/or medically stable with controlled chronic medical conditions (e.g. diabetes mellitus, hypertension ) able to help oneself

Exclusion criteria:

* Known history of systemic hypersensitivity to egg or chicken proteins or any of the vaccine components
* Influenza infection within the past 3 months
* History of Guillain Barre Syndrome (GBS) or brachial neuritis within 6 weeks of previous influenza vaccination
* Treatment with immunosuppressive or other immune-modifying drugs or cancer therapy within the past 6 months
* Any concomitant medication with aspirin
* Participation in other intervention study
* Incapacity to provide fully informed consent or be attentive to follow-up observations resulting from cognitive impairment, abuse of alcohol or drug addiction
* Random blood for Dextrostix more than 200 mg/dL

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Immunological end point | with in 60 days post vaccination
  Vaccine is able to induce a 4-fold rise of Hemagglutination inhibition antibodies 70% of vaccinees within 60 days after vaccination (according to EMA (European Medicines Agency) and CBER (Center for Biologics Evaluation and Research) guidelines)

SECONDARY OUTCOMES:
To assess safety | 60 Days
  To assess safety of the following trivalent inactivated seasonal influenza vaccine in the older age group

OTHER OUTCOMES:
Assess other related immune response | 60 days
  Exploratory objective to assess other related immune response (e.g. anti-neuraminidase)

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Principal Investigator — Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University,, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Boonnak K, Dhitavat J, Thantamnu N, Kosoltanapiwat N, Auayporn M, Jiang L, Puthavathana P, Pitisuttithum P. Immune responses to intradermal and intramuscular inactivated influenza vaccine among older age group. Vaccine. 2017 Dec 19;35(52):7339-7346. doi: 10.1016/j.vaccine.2017.10.106. Epub 2017 Nov 20. PMID 29157960